CLINICAL TRIAL: NCT02582684
Title: A Study to Evaluate Dolutegravir Plus Lamivudine Dual Therapy for the Treatment of Naïve HIV-1-infected Participants
Brief Title: Dolutegravir Plus Lamivudine Dual Therapy in Treatment Naïve HIV-1 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5353; 2UM1AI068636 (NIH)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: DTG 50 mg + 3TC 300 mg (Experimental): Dolutegravir 50mg and Lamivudine 300mg, orally daily
  Interventions: Drug: Dolutegravir; Drug: Lamivudine

INTERVENTIONS:
Drug: Dolutegravir — Participants were prescribed 50 mg of DTG orally daily
  Other Names: DTG
Drug: Lamivudine — Participants were prescribed 300 mg of 3TC orally daily.
  Other Names: 3TC

SUMMARY:
This study was done to see if the combination of two anti-HIV medicines, dolutegravir (DTG, Tivicay) and lamivudine (3TC, Epivir) taken once a day, provide a safe, effective, and well-tolerated treatment for HIV. DTG is a type of HIV medicine called an integrase inhibitor; 3TC is a type of HIV medicine called a reverse transcriptase inhibitor. DTG works by blocking integrase and 3TC works by blocking reverse transcriptase, two HIV proteins (enzymes). This prevents HIV from multiplying and lowers the viral load (amount of HIV in the blood). Both DTG and 3TC are currently part of Food and Drug Administration (FDA) recommended regimens along with a third active drug. Since some HIV medicines have side effects and are costly, there is interest in whether HIV can be successfully controlled with fewer than three HIV drugs.

DETAILED DESCRIPTION:
This study was a phase II, single-arm, open-label pilot study designed to estimate the efficacy of dolutegravir (DTG) plus lamivudine (3TC) as initial combination ART (antiretroviral therapy) in HIV-1 infected treatment naive participants. The target enrollment was 120 participants with a cap of N=90 participants with screening HIV-1 RNA <= 100,000 copies/mL. The study aimed to enroll >= 20% women. The expected follow-up for each participant was 52 weeks.

Visits occurred at screening, entry, and weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52 from study entry. All signs/symptoms within 30 days prior to entry were recorded. Subsequently, grade 2 or higher rash and all other grade 3 or higher signs and symptoms were recorded. All participants underwent routine monitoring including plasma HIV-1 RNA levels, CD4+ cell count, hematology, chemistry, urinalysis, and pregnancy testing (for women of reproductive potential).

Population-based protease (PR), reverse transcriptase (RT) and integrase genotyping were done at the time of confirmed virologic failure. Plasma samples were stored for potential future studies to assess the impact of adherence, drug-resistant minority viral variants, and DTG exposure on virologic and CD4+ cell count responses to DTG plus 3TC. All participants also underwent UGT1A1 genotyping.

ELIGIBILITY:
NOTE: Further information on the eligibility criteria can be found in the study protocol.

Inclusion Criteria:

* HIV-1 infection.
* Plasma HIV-1 RNA ≥1000 copies/mL and <500,000 copies/mL obtained within 90 days prior to study entry.
* No evidence of any RT, any integrase, or major protease resistance mutation (according to the 2014 IAS-USA drug resistance mutations list, available at https://www.iasusa.org/sites/default/files/tam/22-3-642.pdf) based on pre-ARV (antiretroviral) treatment genotype performed any time prior to study entry.
* ARV treatment drug-naive (defined as no previous ARV treatment at any time prior to study entry, with the exception of successful post-exposure prophylaxis (PEP) or pre-exposure prophylaxis (PrEP).
* The following laboratory values obtained within 45 days prior to study entry:

  * ANC (absolute neutrophil count) ≥750/mm^3
  * Hemoglobin ≥10.0 g/dL
  * Platelets ≥ 50,000/mm^3
  * Calculated creatinine clearance (CrCl) ≥50 mL/min, as estimated by the Cockcroft-Gault equation
  * AST (aspartate aminotransferase) <5 x ULN (upper limit of normal)
  * ALT (alanine aminotransferase) <5x ULN
  * Total bilirubin <1.5 x ULN
* Hepatitis B surface antigen negative within 45 days prior to study entry.
* For women with reproductive potential, negative serum or urine pregnancy test at screening and within 48 hours prior to study entry.
* If participating in sexual activity that could lead to pregnancy, female participants with reproductive potential must have agreed to use one form of contraceptive as listed in the protocol while receiving protocol-specified medications and for 30 days after stopping the medications.
* Ability and willingness of participant or legal representative to provide informed consent.

Exclusion Criteria:

* Serious illness requiring systemic treatment and/or hospitalization.
* Treatment within 30 days prior to study entry with immune modulators such as systemic steroids, interleukins, interferons, granulocyte colony-stimulating factor (G-CSF), erythropoietin, or any investigational therapy.
* Pregnancy or breastfeeding.
* Receipt of systemic cytotoxic chemotherapy or dofetilide.
* Known allergy/sensitivity to any of the study drugs or their formulations.
* Active drug or alcohol use or dependence that may interfere with adherence to study requirements, in the opinion of the site investigator.
* Active hepatitis C virus (HCV) treatment or anticipated need for treatment within study period.
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Severe hepatic impairment (Class C) as determined by Child-Pugh classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Gulick, MD, MPH, Study Chair — Weill Medical College of Cornell University; Babafemi Taiwo, MBBS, Study Chair — Northwestern University
Locations (26):
- United States (25):
  - University of Southern California CRS (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Univ. of Miami AIDS CRS (901), Miami, Florida
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - Cornell CRS (7804), New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU -Chelsea (7803), New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - 3201 Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - The Miriam Hospital ACTG CRS (2951), Providence, Rhode Island
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - 31443 Trinity Health and Wellness Center CRS, Dallas, Texas
  - Houston AIDS Research Team CRS (31473), Houston, Texas
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Derived] Nyaku AN, Zheng L, Gulick RM, Olefsky M, Berzins B, Wallis CL, Godfrey C, Sax PE, Acosta EP, Haas DW, Smith KY, Sha BE, Van Dam CN, Taiwo BO; ACTG A5353 Study Team. Dolutegravir plus lamivudine for initial treatment of HIV-1-infected participants with HIV-1 RNA <500 000 copies/mL: week 48 outcomes from ACTG 5353. J Antimicrob Chemother. 2019 May 1;74(5):1376-1380. doi: 10.1093/jac/dky564. PMID 30668695
- [Derived] Taiwo BO, Zheng L, Stefanescu A, Nyaku A, Bezins B, Wallis CL, Godfrey C, Sax PE, Acosta E, Haas D, Smith KY, Sha B, Van Dam C, Gulick RM. ACTG A5353: A Pilot Study of Dolutegravir Plus Lamivudine for Initial Treatment of Human Immunodeficiency Virus-1 (HIV-1)-infected Participants With HIV-1 RNA <500000 Copies/mL. Clin Infect Dis. 2018 May 17;66(11):1689-1697. doi: 10.1093/cid/cix1083. PMID 29253097
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf?sfvrsn=8
- See also: FDA Snapshot Definition (refer to Appendix A in FDA Snapshot PDF) — https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm355128.pdf
- See also: DAIDS Adverse Events Manual, Version 2.0 January 2010 — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 122 participants were accrued.
Period: Overall Study
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Started | 122
Completed | 105
Not Completed | 17
Not completed — Unable to contact subject/parent | 4
Not completed — Subject not able to get to clinic | 10
Not completed — Subject withdrew consent | 1
Not completed — Found to be ineligible after enrollment | 2

BASELINE CHARACTERISTICS:
Population: All eligible participants enrolled.
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
Age, Continuous [Median (Inter-Quartile Range); unit: Years]
  Age | 30 [24 to 41]
Age, Customized [Count of Participants; unit: Participants]
  Age Category: 18-29 years | 58
  Age Category: 30-39 years | 29
  Age Category: 40-49 years | 17
  Age Category: 50-59 years | 12
  Age Category: >= 60 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 34
  Race/Ethnicity: Black Non-Hispanic | 48
  Race/Ethnicity: Hispanic (Regardless of Race) | 32
  Race/Ethnicity: Asian, Pacific Islander | 2
  Race/Ethnicity: More than one race | 2
  Race/Ethnicity: Does not want to report | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 3
  United States | 117
Intravenous Drug Use [Count of Participants; unit: Participants]
  Never | 113
  Currently | 2
  Previously | 5
CD4 Count, Continuous [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: 2 participants with missing baseline CD4 counts.
  cells/mm^3
    number analyzed (Participants) | 118
    (all) | 387 [288 to 596]
CD4 Count, Categorized [Count of Participants; unit: Participants]
  <200 cells/mm^3 | 16
  200-349 cells/mm^3 | 27
  350-499 cells/mm^3 | 30
  500-649 cells/mm^3 | 19
  650-799 cells/mm^3 | 15
  >=800 cells/mm^3 | 11
  Missing | 2
CD8 Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Total of 13 participants missing CD8 Count at baseline.
  cells/mm^3
    number analyzed (Participants) | 107
    (all) | 871 [610 to 1167]
CD4/CD8 Ratio [Median (Inter-Quartile Range); unit: ratio] — Population: Total of 13 participants had missing measurements that contribute to the CD4/CD8 ratio.
  ratio
    number analyzed (Participants) | 107
    (all) | 0.44 [0.31 to 0.70]
Screening HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 4.70 [4.08 to 5.00]
Baseline HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] — Baseline HIV-1 RNA is defined as the last nonmissing observation on or prior to first dose date after screening.
  log10 copies/mL | 4.61 [3.94 to 5.05]
Baseline HIV-1 RNA Category [Count of Participants; unit: Participants] — Baseline HIV-1 RNA is defined as the last nonmissing observation on or prior to first dose date after screening.
  Participants
    < 1,000 copies/mL | 1
    1,000 - 9,999 copies/mL | 34
    10,000 - 99,999 copies/mL | 48
    100,000 - 200,000 copies/mL | 23
    > 200,000 copies/mL | 14
Hepatitis C Antibody Status [Count of Participants; unit: Participants]
  Positive | 4
  Negative | 116
Post-exposure Prophylaxis or Pre-Exposure Prophylaxis History [Count of Participants; unit: Participants]
  Yes | 1
  No | 119

OUTCOME MEASURES:

1. Primary Outcome: Virologic Status at Week 24
Description: Numbers of Participants With Virologic Success, Virologic Non-Success, and no Virologic Data at Week 24 Window are provided below.
  Virologic success is defined as HIV-1 RNA <50 copies/mL and on study treatment (FDA Snapshot definition).
Time Frame: At 24 weeks after study entry
Population: All eligible participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
Participants
  Virologic success | 108
  Virologic non-success | 5
  No virologic data in window | 7
Statistical Analysis 1: Comparison: Arm 1: DTG 50 MG + 3TC 300 mg; Test type: Other — Binomial Proportion of Participants with Virologic Success and 95% Confidence Interval; proportion = 0.90, 95% CI 2-sided [0.83 to 0.95] — Confidence interval was calculated using the Clopper-Pearson exact method

2. Secondary Outcome: Virologic Status at Week 12
Description: Numbers of Participants With Virologic Success, Virologic Non-Success, and no Virologic Data at Week 12 Window are provided below.
  Virologic success is defined as HIV-1 RNA <50 copies/mL and on study treatment (FDA Snapshot definition).
Time Frame: At 12 weeks after study entry
Population: All eligible participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
Participants
  Virologic success | 107
  Virologic non-success | 7
  No virologic data in window | 6
Statistical Analysis 1: Comparison: Arm 1: DTG 50 MG + 3TC 300 mg; Test type: Other — Binomial Proportion of Participants with Virologic Success and 95% Confidence Interval; Proportion = 0.89, 95% CI 2-sided [0.82 to 0.94] — Confidence interval was calculated using the Clopper-Pearson exact method

3. Secondary Outcome: Virologic Status at Week 48
Description: Numbers of Participants With Virologic Success, Virologic Non-Success, and no Virologic Data at Week 48 Window are provided below.
  Virologic success is defined as HIV-1 RNA <50 copies/mL and on study treatment (FDA Snapshot definition).
Time Frame: At 48 weeks after study entry
Population: All eligible participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
Participants
  Virologic success | 102
  Virologic non-success | 6
  No virologic data in window | 12
Statistical Analysis 1: Comparison: Arm 1: DTG 50 MG + 3TC 300 mg; Test type: Other — Binomial Proportion of Participants with Virologic Success and 95% Confidence Interval; proportion = 0.85, 95% CI 2-sided [0.77 to 0.91] — Confidence interval was calculated using the Clopper-Pearson exact method

4. Secondary Outcome: Virologic Failure
Description: Virologic failure is defined as follows:
  * Weeks 16 or 20: confirmed plasma HIV-1 RNA > 400 copies/mL
  * Week 24 or later: confirmed plasma HIV-1 RNA > 200 copies/mL
    1. Participants were evaluated for virologic failure regardless of whether on study treatment.
    2. Confirmation was determined based on any two consecutive evaluations meeting the virologic failure definition regardless of the time between them.
    3. Participants discontinuing the study (for any reason, including death and lost to follow-up) were considered virologic failures if their last measurement met the definition of virologic failure but no confirmatory measurement was obtained. All other participants' follow-up was censored immediately after the last available plasma HIV-1 RNA measurement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: All eligible participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
Participants
  Yes | 4
  No | 116

5. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA < 50 Copies/mL - Missing = Failure
Description: Proportion of participants with HIV-1 RNA < 50 copies/mL by week, ITT (Intention To Treat; missing/off study/off treatment = failure) population.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: The population here is the ITT (missing/off study/off treatment = failure) population. The numerator includes participants with HIV-1 RNA < 50 copies/mL and still on initial treatment; the denominator includes all participants with potential for the given week of follow-up based on the date of registration.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
proportion of participants
  Week 2 | 0.40 [0.31 to 0.49]
  Week 4 | 0.68 [0.58 to 0.76]
  Week 8 | 0.85 [0.77 to 0.91]
  Week 12 | 0.89 [0.82 to 0.94]
  Week 16 | 0.88 [0.80 to 0.93]
  Week 20 | 0.90 [0.83 to 0.95]
  Week 24 | 0.90 [0.83 to 0.95]
  Week 32 | 0.88 [0.80 to 0.93]
  Week 40 | 0.89 [0.82 to 0.94]
  Week 48 | 0.84 [0.76 to 0.90]

6. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA < 200 Copies/mL - Missing = Failure
Description: Proportion of participants with HIV-1 RNA < 200 copies/mL by week, ITT (missing/off study/off treatment = failure) population.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: The population here is the ITT (missing/off study/off treatment = failure) population. The numerator includes participants with HIV-1 RNA < 200 copies/mL and still on initial treatment; the denominator includes all participants with potential for the given week of follow-up based on the date of registration.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
proportion of participants
  Week 2 | 0.68 [0.59 to 0.77]
  Week 4 | 0.90 [0.83 to 0.95]
  Week 8 | 0.95 [0.89 to 0.98]
  Week 12 | 0.93 [0.87 to 0.97]
  Week 16 | 0.92 [0.85 to 0.96]
  Week 20 | 0.95 [0.89 to 0.98]
  Week 24 | 0.92 [0.85 to 0.96]
  Week 32 | 0.89 [0.82 to 0.94]
  Week 40 | 0.91 [0.84 to 0.95]
  Week 48 | 0.87 [0.79 to 0.92]

7. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA <50 Copies/mL - Missing = Ignored
Description: Proportion of participants with HIV-1 RNA < 50 copies/mL by week, ITT (missing = ignored) population.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: ITT Missing = Ignored. The numerator includes participants with HIV-1 RNA < 50 copies/mL; the denominator includes all participants with an HIV-1 RNA evaluation at the given week.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
proportion of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 0.41 [0.32 to 0.51]
  Week 4: number analyzed (Participants) | 115
  Week 4 | 0.70 [0.61 to 0.79]
  Week 8: number analyzed (Participants) | 116
  Week 8 | 0.88 [0.81 to 0.93]
  Week 12: number analyzed (Participants) | 114
  Week 12 | 0.94 [0.88 to 0.97]
  Week 16: number analyzed (Participants) | 112
  Week 16 | 0.94 [0.88 to 0.97]
  Week 20: number analyzed (Participants) | 115
  Week 20 | 0.94 [0.88 to 0.98]
  Week 24: number analyzed (Participants) | 114
  Week 24 | 0.96 [0.90 to 0.99]
  Week 32: number analyzed (Participants) | 113
  Week 32 | 0.93 [0.87 to 0.97]
  Week 40: number analyzed (Participants) | 114
  Week 40 | 0.95 [0.89 to 0.98]
  Week 48: number analyzed (Participants) | 109
  Week 48 | 0.94 [0.87 to 0.97]

8. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA <200 Copies/mL- ITT Missing = Ignored
Description: Proportion of participants with HIV-1 RNA < 200 copies/mL by week, ITT (missing = ignored) population.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: ITT Missing = Ignored. The numerator includes participants with HIV-1 RNA < 200 copies/mL; the denominator includes all participants with an HIV-1 RNA evaluation at the given week.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
proportion of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 0.71 [0.62 to 0.79]
  Week 4: number analyzed (Participants) | 115
  Week 4 | 0.94 [0.88 to 0.98]
  Week 8: number analyzed (Participants) | 116
  Week 8 | 0.98 [0.94 to 1.00]
  Week 12: number analyzed (Participants) | 114
  Week 12 | 0.98 [0.94 to 1.00]
  Week 16: number analyzed (Participants) | 112
  Week 16 | 0.98 [0.94 to 1.00]
  Week 20: number analyzed (Participants) | 115
  Week 20 | 0.99 [0.95 to 1.00]
  Week 24: number analyzed (Participants) | 114
  Week 24 | 0.97 [0.93 to 0.99]
  Week 32: number analyzed (Participants) | 113
  Week 32 | 0.95 [0.89 to 0.98]
  Week 40: number analyzed (Participants) | 114
  Week 40 | 0.96 [0.91 to 0.99]
  Week 48: number analyzed (Participants) | 109
  Week 48 | 0.96 [0.91 to 0.99]

9. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA <50 Copies/mL- As Treated
Description: Proportion of participants with HIV-1 RNA < 50 copies/mL by week, as treated population.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: As Treated: purely virologic missing = ignored. The numerator includes participants with HIV-1 RNA < 50 copies/mL and still on initial treatment; the denominator includes participants on initial treatment with an HIV-1 RNA evaluation at the given week.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
proportion of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 0.41 [0.32 to 0.51]
  Week 4: number analyzed (Participants) | 115
  Week 4 | 0.70 [0.61 to 0.79]
  Week 8: number analyzed (Participants) | 116
  Week 8 | 0.88 [0.81 to 0.93]
  Week 12: number analyzed (Participants) | 114
  Week 12 | 0.94 [0.88 to 0.97]
  Week 16: number analyzed (Participants) | 112
  Week 16 | 0.94 [0.88 to 0.97]
  Week 20: number analyzed (Participants) | 115
  Week 20 | 0.94 [0.88 to 0.98]
  Week 24: number analyzed (Participants) | 112
  Week 24 | 0.96 [0.91 to 0.99]
  Week 32: number analyzed (Participants) | 110
  Week 32 | 0.95 [0.90 to 0.99]
  Week 40: number analyzed (Participants) | 110
  Week 40 | 0.97 [0.92 to 0.99]
  Week 48: number analyzed (Participants) | 104
  Week 48 | 0.97 [0.92 to 0.99]

10. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA <200 Copies/mL- As Treated
Description: Proportion of participants with HIV-1 RNA < 200 copies/mL by week, as treated population.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: As Treated: purely virologic missing=ignored. The numerator includes participants with HIV-1 RNA < 200 copies/mL and still on initial treatment; the denominator includes participants on initial treatment with an HIV-1 RNA evaluation at the given week.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
proportion of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 0.71 [0.62 to 0.79]
  Week 4: number analyzed (Participants) | 115
  Week 4 | 0.94 [0.88 to 0.98]
  Week 8: number analyzed (Participants) | 116
  Week 8 | 0.98 [0.94 to 1.00]
  Week 12: number analyzed (Participants) | 114
  Week 12 | 0.98 [0.94 to 1.00]
  Week 16: number analyzed (Participants) | 112
  Week 16 | 0.98 [0.94 to 1.00]
  Week 20: number analyzed (Participants) | 115
  Week 20 | 0.99 [0.95 to 1.00]
  Week 24: number analyzed (Participants) | 112
  Week 24 | 0.98 [0.94 to 1.00]
  Week 32: number analyzed (Participants) | 110
  Week 32 | 0.97 [0.92 to 0.99]
  Week 40: number analyzed (Participants) | 110
  Week 40 | 0.99 [0.95 to 1.00]
  Week 48: number analyzed (Participants) | 104
  Week 48 | 1.00 [0.97 to 1.00]

11. Secondary Outcome: CD4+ Cell Count
Description: CD4+ cell counts by study week.
Time Frame: Baseline, weeks 4, 12, 24, and 48
Population: All eligible participants enrolled with CD4 count results available at a given visit.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
cells/mm^3
  Week 0: number analyzed (Participants) | 118
  Week 0 | 387 [288 to 596]
  Week 4: number analyzed (Participants) | 118
  Week 4 | 473 [358 to 727]
  Week 12: number analyzed (Participants) | 115
  Week 12 | 520 [395 to 783]
  Week 24: number analyzed (Participants) | 115
  Week 24 | 582 [416 to 871]
  Week 48: number analyzed (Participants) | 107
  Week 48 | 579 [451 to 830]

12. Secondary Outcome: Change in CD4+ Cell Count
Description: Change in CD4+ cell counts by study week. Change was calculated as value at the later visit minus the value at baseline.
Time Frame: Baseline, weeks 4, 12, 24, and 48
Population: All eligible participants enrolled with CD4 cell count results available at baseline and the given visit.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
cells/mm^3
  Change from Baseline to Week 4: number analyzed (Participants) | 116
  Change from Baseline to Week 4 | 78 [10 to 154]
  Change from Baseline to Week 12: number analyzed (Participants) | 113
  Change from Baseline to Week 12 | 122 [67 to 185]
  Change from Baseline to Week 24: number analyzed (Participants) | 113
  Change from Baseline to Week 24 | 167 [86 to 275]
  Change from Baseline to Week 48: number analyzed (Participants) | 105
  Change from Baseline to Week 48 | 182 [104 to 284]

13. Secondary Outcome: Number of HIV-1 Drug Resistance Mutation Occurrences in Participants
Description: Number of HIV-1 drug resistance mutation occurrences participants with virologic failure and FDA snapshot non-successes. Participants that had one drug class resistance mutation may have one or more mutations.
Time Frame: at the time of virologic failure
Population: Of the enrolled eligible participants, those with virologic failures had resistance testing done.
Measure: Number; unit: number of mutation occurrences
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 4
number of mutation occurrences
  NRTI mutation | 1
  NNRTI mutation | 1
  INI mutation | 1

14. Secondary Outcome: Fasting Lipids and Glucose
Description: Fasting lipids include: total cholesterol, triglycerides, LDL cholesterol, HDL cholesterol, and glucose. Fasting was set to be 8 hours prior to the sample collection.
Time Frame: Baseline and week 48
Population: All eligible participants enrolled with lipids results available at a given time point.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
mg/dL
  Baseline Total Cholesterol: number analyzed (Participants) | 92
  Baseline Total Cholesterol | 151 [123 to 171]
  Week 48 Total Cholesterol: number analyzed (Participants) | 100
  Week 48 Total Cholesterol | 154 [136 to 189]
  Baseline LDL Cholesterol: number analyzed (Participants) | 91
  Baseline LDL Cholesterol | 85 [69 to 107]
  Week 48 LDL Cholesterol: number analyzed (Participants) | 99
  Week 48 LDL Cholesterol | 86 [69 to 117]
  Baseline HDL Cholesterol: number analyzed (Participants) | 92
  Baseline HDL Cholesterol | 39 [33 to 49]
  Week 48 HDL Cholesterol: number analyzed (Participants) | 100
  Week 48 HDL Cholesterol | 46 [38 to 56]
  Baseline Triglycerides: number analyzed (Participants) | 92
  Baseline Triglycerides | 91 [70 to 133]
  Week 48 Triglycerides: number analyzed (Participants) | 100
  Week 48 Triglycerides | 98 [60 to 150]
  Baseline Glucose: number analyzed (Participants) | 96
  Baseline Glucose | 84 [78 to 92]
  Week 48 Glucose: number analyzed (Participants) | 62
  Week 48 Glucose | 86 [81 to 93]

15. Secondary Outcome: Creatinine Clearance
Description: Creatinine clearance was estimated by the Cockcroft-Gault equation.
Time Frame: Baseline, weeks 4, 12, 24, 32, 40 and 48
Population: All eligible participants enrolled with creatinine clearance results available at a given time point.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
mL/min
  Week 0 | 126.0 [106.8 to 139.9]
  Week 4: number analyzed (Participants) | 116
  Week 4 | 112.9 [96.6 to 133.2]
  Week 12: number analyzed (Participants) | 114
  Week 12 | 112.0 [97.8 to 133.3]
  Week 24: number analyzed (Participants) | 114
  Week 24 | 114.7 [96.8 to 132.7]
  Week 32: number analyzed (Participants) | 111
  Week 32 | 115.5 [97.1 to 138.6]
  Week 40: number analyzed (Participants) | 113
  Week 40 | 112.7 [97.4 to 138.7]
  Week 48: number analyzed (Participants) | 111
  Week 48 | 114.4 [101.2 to 133.5]

16. Secondary Outcome: Number of Participants With Grade 3 of Higher Adverse Events
Description: Number of participants who experienced an AE (sign/symptom or laboratory abnormality) of Grade 3 or higher. The AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (see reference in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening.
Time Frame: from study treatment dispensation through up to week 52 or until study discontinuation
Population: All eligible participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
Number analyzed (Participants) | 120
Participants | 16

ADVERSE EVENTS:
Time Frame: From study entry through up to week 52 or until study discontinuation
Description: The protocol required reporting of all diagnoses (identified by the ACTG criteria for clinical events and other diseases), signs/symptoms and laboratory values of >= Grade 3 and events that led to a change in treatment or that met ICH, EAE, or SAE guidelines, regardless of grade. Creatinine and creatinine clearance were reported regardless of grade. The DAIDS AE Grading Table (Version 2.0) and Expedited AE Manual (Version 2.0) were used.
Arm/Group | Arm 1: DTG 50 MG + 3TC 300 mg
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 3/122
Other Adverse Events (participants affected / at risk) | 75/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: DTG 50 MG + 3TC 300 mg (N=122)
Suicidal ideation (Psychiatric disorders) | 3
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: DTG 50 MG + 3TC 300 mg (N=122)
Urethritis gonococcal (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 10
Blood cholesterol increased (Investigations) | 20
Blood creatinine abnormal (Investigations) | 10
Blood glucose increased (Investigations) | 11
Blood sodium decreased (Investigations) | 7
Blood triglycerides increased (Investigations) | 30
Low density lipoprotein increased (Investigations) | 19
Neutrophil count decreased (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02582684/SAP_000.pdf
  • Study Protocol (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT02582684/Prot_001.pdf